CLINICAL TRIAL: NCT06059443
Title: mLab App Plus: A Randomized Controlled Trial of an mHealth Intervention for Increasing Access to HIV and Syphilis Testing and Care Among Young Men
Brief Title: mLab App Plus: A Randomized Controlled Trial of a Mobile Health (mHealth) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Professor of Disease Prevention and Health Promotion (Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAU3380; K24NR018621 (NIH); R01MH118151 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections; Sexually Transmitted Diseases, Viral; Syphilis
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases, Viral; Syphilis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of two trial arms using the randomization module in REDCap. We will use block randomization with randomly permutated blocks to reduce opportunities for selection bias
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mLab App Plus (Experimental): Participants randomized to intervention will receive standard of care counseling, complete online surveys, be provided with the mLab App Plus, and a box of condoms. The intervention arm will also complete two HIV/Syphilis Ab Combo Rapid Tests (DPP® HIV-Syphilis Test) at their baseline (first test) and 3-month follow- up (second test) appointments.
  Interventions: Behavioral: mLab App Plus
- Standard of Care (No Intervention): Participants randomized to standard care will receive standard of care counseling, complete online surveys and be sent an email with links to mobile-optimized online prevention information, including Pre-Exposure Prophylaxis(PrEP) and HIV/STI testing information found on the Centers for Disease Control (CDC) website, and a box of condoms.

INTERVENTIONS:
Behavioral: mLab App Plus — Participants will use the mLab Plus app to test for Syphilis and HIV using the DPP HIV/Syphilis Test
  Arms: mLab App Plus

SUMMARY:
Men who have sex with men (MSM), especially young men who have sex with men (YMSM), and transgender women (TGW) have some of the highest rates of HIV and syphilis diagnoses in the United States. The goal of this study is to pilot the mobile Lab (mLab) App Plus to assess YMSM's and YTGW's abilities to perform and interpret self-tests for HIV and syphilis and consequently increase the number of YMSM and young transgender woman (YTGW) who initiate self-testing for HIV and syphilis.

DETAILED DESCRIPTION:
From 2018 to 2019, the rate of syphilis increased by 11.2%. It has increased steadily since 2000 especially among men, in which MSM bear a disproportionate majority of cases (47% of all cases were among MSM in 2019). HIV and syphilis rates continue to rise among YMSM. While MSM account for only about 2% of the US population, they are most affected by HIV, constituting 56% of people living with HIV (PLWH).

Moreover, the rate of syphilis among MSM is profoundly elevated, at least 100 times higher than that in men who have sex with women and even higher among YMSM. Importantly, syphilis makes it easier to both acquire and transmit HIV, and about half of MSM who have syphilis are co-infected with HIV. The risk of syphilis and HIV continues to rise in YMSM in New York City, the study site. Given these epidemiologic risk factors for HIV and syphilis, there is a strong scientific premise for this pilot study that proposes to test innovative and effective HIV and sexually transmitted infection (STI) testing, prevention, and treatment models. Given that approximately 17% of MSM living with HIV in the U.S. are unaware of their status and significant comorbid syphilis in that population, both pathogens may be simultaneously transmitted. The increasing number of syphilis diagnosed in MSM highlights the importance of STI control in this population, not just for the health of the patient, but also for prevention of HIV and syphilis in uninfected persons. YMSM and YTGW, and specifically Blacks and Latinos, are disproportionately infected with HIV.

In response to the need for interventions to increase HIV testing in youth, our study team developed the mLab App, which affords advantages over existing self-test options to support the potential for higher uptake of the HIV self-test. The app provides HIV prevention information, push notification reminders for testing, step-by-step instructions for using the OraQuick HIV tests (OraQuick), and an image upload function so individuals can send an image of their OraQuick HIV test to the study team. In response to the mLab App study and the scientific evidence of need for at-home syphilis point of care (POC) testing among YMSM and YTGW, we propose to implement the mLab App Plus to assess YMSM's and YTGW's abilities to perform and interpret self-tests for HIV and syphilis and consequently increase the number of YMSM and YTGW who initiate self-testing for HIV and syphilis.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years of age
* Assigned male sex at birth and identify as (1) a man or (2) a trans woman
* Understand and read English
* Self-identify as any race or ethnicity
* Substantial risk for acquiring HIV infection per CDC (Centers for Disease Control) guidance
* All participants must report having sex with a man/men
* Smart phone ownership
* Self-report being HIV-negative or unknown status
* Self-report being negative for syphilis or unknown status
* Not having been tested for HIV or syphilis in the past 3 months
* Understand the limitations of the duplex lateral flow test and the mLab App Plus (e.g., a confirmatory test is needed and self-test must be performed in the presence of a qualified clinician)

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Assigned male sex at birth and identify as (1) a man or (2) a trans woman
Enrollment: 40 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Vanderbilt University, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Participants randomized to standard care will receive standard of care counseling, complete online surveys and be sent an email with links to mobile-optimized online prevention information, including Pre-Exposure Prophylaxis(PrEP) and HIV/sexually transmitted infection (STI) testing information found on the Centers for Disease Control (CDC) website, and a box of condoms.
Period: Overall Study
Arm/Group | mLab App Plus | Standard of Care
Started | 20 | 20
Completed | 16 | 18
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mLab App Plus | Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.33 (3.94) | 28.71 (4.99) | 28.52 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 5 | 4 | 9
  Race: White | 8 | 8 | 16
  Race: Asian | 5 | 2 | 7
  Race: Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Race: Unknown | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
The Number of Participants Who Are Able to Self-administer the DPP® HIV-Syphilis Test With mLab App [Count of Participants; unit: Participants] — A successful self-test is defined as having completed the DPP® HIV-Syphilis test by themselves and having accurately identified and interpreted their HIV and Syphilis statuses as determined by the supervising clinician. In the event that the clinician, rather than the participant administers the DPP® HIV-Syphilis test, the test is not recorded as a successful self-test. Population: The Standard of Care Arm did not test with mLab App Plus
  Participants
    number analyzed (Participants) | 20 | 0 | 20
    (all) | 16 |  | 16
The Number of Negative/Positive Results [Count of Participants; unit: Participants] — The number of participants who tested reactive (R) or positive and/or non-reactive (NR) or negative for syphilis and HIV using the DPP® HIV-Syphilis test with mLab App Plus. Test results appear in a single reading with the results of both HIV and syphilis. Population: Zero analyzed in the Standard of Care (SOC) Arm, as the SOC Arm did not use the mLab Ap Plus.
  Participants
    Negative (HIV)/ Negative (Syphilis): number analyzed (Participants) | 20 | 0 | 20
    Negative (HIV)/ Negative (Syphilis) | 15 |  | 15
    Negative (HIV)/ Positive (Syphilis): number analyzed (Participants) | 20 | 0 | 20
    Negative (HIV)/ Positive (Syphilis) | 3 |  | 3
    Positive (HIV)/ Negative (Syphilis): number analyzed (Participants) | 20 | 0 | 20
    Positive (HIV)/ Negative (Syphilis) | 1 |  | 1
    Positive (HIV)/ Positive (Syphilis): number analyzed (Participants) | 20 | 0 | 20
    Positive (HIV)/ Positive (Syphilis) | 1 |  | 1
Number of Participants referred for HIV/STI Services [Count of Participants; unit: Participants] — Using the count of referral for participants that tested positive (reactive) to HIV and/or syphilis using mLabApp Plus. Population: 5 analyzed as 5 participants tested positive for HIV/Syphilis. Zero analyzed in the Standard of Care (SOC) Arm, as the SOC Arm did not use the mLab App Plus.
  Participants
    number analyzed (Participants) | 5 | 0 | 5
    (all) | 5 |  | 5
Number of Participants Linked to HIV/STI Prevention or Care Services [Count of Participants; unit: Participants] — The number of participants linked to and that attend one appointment for HIV/STI services. Population: 5 analyzed as 5 participants tested positive for HIV/Syphilis. Zero analyzed in the Standard of Care (SOC) Arm, as the SOC Arm did not use the mLab App Plus.
  Participants
    number analyzed (Participants) | 5 | 0 | 5
    (all) | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Are Able to Self-administer the DPP® HIV-Syphilis Test With mLab App Plus
Description: A successful self-test is defined as having completed the DPP® HIV-Syphilis test by themselves and having accurately identified and interpreted their HIV and Syphilis statuses as determined by the supervising clinician. In the event that the clinician, rather than the participant administers the DPP® HIV-Syphilis test, the test is not recorded as a successful self-test.
Time Frame: 3-Month Follow-up
Population: The Standard of Care arm did not receive access to the mLab App Plus.
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Plus
Number analyzed (Participants) | 20
Participants | 12

2. Secondary Outcome: The Number of Negative/Positive Results
Description: The number of participants who tested reactive (R) or positive and/or non-reactive (NR) or negative for syphilis and HIV using the DPP® HIV-Syphilis test with mLab App Plus. Test results appear in a single reading with the results of both HIV and syphilis.
Time Frame: 3-Month Follow-up
Population: 15 participants analyzed in the mLab App Plus arm as data was collected from 15 out of 20 (n=4 did not complete the 3-month follow up and a sample was not collected for n=1). The Standard of Care arm did not receive access to the mLab App Plus.
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Plus
Number analyzed (Participants) | 15
Participants
  Negative (HIV) / Negative (Syphilis) | 12
  Negative (HIV) / Positive (Syphilis) | 3
  Positive (HIV) / Negative (Syphilis) | 0
  Positive (HIV) /Positive (Syphilis) | 0

3. Secondary Outcome: Number of Participants Referred for HIV/STI Services (Participants With HIV and/or Syphilis Only)
Description: The number of Young Men who have sex with men/ Young transgender women referred for HIV/STI services (participants with HIV and/or syphilis only). Using count of referral for participants that tested positive (reactive) to HIV and/or syphilis using mLabApp Plus.
Time Frame: 3-Month Follow-up
Population: Three analyzed as three tested positive using the mLabApp Plus. The Standard of Care arm did not receive access to the mLab App Plus.
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Plus
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Number of Participants Linked to (Attend One Appointment) HIV/STI Prevention or Care Services
Description: The number of Young Men who have sex with men/ Young transgender women linked to (attend one appointment) HIV/STI prevention or care services. Using count of appointments attended.
Time Frame: 3-Month Follow-up
Population: Three analyzed as three participants tested positive at month 3
Measure: Count of Participants; unit: Participants
Arm/Group | mLab App Plus
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | mLab App Plus | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT06059443/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT06059443/ICF_001.pdf